CLINICAL TRIAL: NCT02905786
Title: Implementation of a Multifaceted Intervention to Optimize Care for Heart Failure Patients in Primary Care: Protocol of a Pilot Study
Brief Title: Protocol of a Pilot Study to Optimize Care for Heart Failure Patients in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Miek Smeets, PhD student, KU Leuven
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S59579
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure
Keywords: General Practice; Nurse practitioner; Natriuretic peptides; Clinical audit
MeSH Terms: conditions — Heart Failure | interventions — Clinical Audit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cobas h232 (Roche Diagnostics) — NT-proBNP point-of-care test
Other: Clinical audit and feedback — Clinical audit and feedback to detect previously unrecognized HF patients and inform GPs about their current quality of HF care
Other: Assistance by a specialized HF nurse — Assistance by a specialized HF nurse in general practice for education of patients, advice in diagnosis and treatment, transition of care

SUMMARY:
Heart failure (HF) imposes a burden for patients and health economics. Although guidelines exist, they are not implemented as such in the Belgian health care system. General practitioners (GPs) are confronted with the broadest range of HF management. Therefore, a multifaceted intervention will be implemented in Belgian general practice to support GPs in the implementation of evidence-based HF guidelines. This multifaceted intervention will consist of audit and feedback as a method to detect unrecognized HF patients and increase awareness for proactive HF management. Additionally, a NT-proBNP point-of-care test will be offered to every practice to improve detection and adequate diagnosis of HF patients. Furthermore, a specialist HF nurse will assist GPs in education of patients, optimization of treatment and transition of care. The investigators' aim is evaluating the feasibility of the implementation of this multifaceted intervention in general practice and the evolution in predefined quality indicators.

DETAILED DESCRIPTION:
Objectives:

The objective of this pilot study is to assess the feasibility of a multifaceted intervention to optimize care for HF patients in Belgian general practice. It is not a primary objective to study the effectiveness of the intervention on the defined outcomes, since follow-up might be too short, however the evolution in quality will be evaluated. Specific research questions are:

1. Do general practitioners use the NT-proBNP POC test and how does it influence practice?
2. Do general practitioners use the assistance of the HF nurse and how does it influence practice?
3. Does this intervention improve quality of care for HF patients in primary care?
4. Does this intervention improve quality of life for HF patients in primary care?
5. Is this intervention/data collection method feasible? How do participating GPs and investigators experience the interventions?

Data collection:

* Measurements at baseline and after 6 months of follow-up
* Baseline demographic data on patient age, gender, years since the diagnosis of HF, cardiovascular comorbidities (hypertension, ischemic heart disease, valvular heart disease, atrial fibrillation, cerebrovascular disease, peripheral arterial disease), non-cardiovascular comorbidities (diabetes, depression, chronic obstructive pulmonary disease, dementia), the last two blood pressure measurements, last 2 creatinine measurements and the last two values of the estimated glomerular filtration rate (eGFR), last date of GP consultation, involvement of cardiologist (yes/no), last date of cardiologist appointment, echocardiography (yes/no), last date of echocardiography report, ejection fraction (EF), diastolic dysfunction (yes/no), clinically relevant valvular dysfunction (yes/no), left ventricular hypertrophy (yes/no), left atrial enlargement (yes/no) and heart failure treatment with dosage (diuretics, ACE-I, ARB, B-blockers, MRA, digoxin) will be collected. Additionally, the number of chronic medications and the number of chronic comorbidities will be collected. Furthermore, the MLHF-Q will be collected to evaluate patients' quality of life and grip strength (only at baseline) as a predictor of functional decline, disability and mortality. At baseline, HF hospitalization during the last three years will be registered based on discharge letters in the EHR. All hospitalizations and mortality will be collected at practice level during the study course. Data on physician age, gender, years of experience and practice organization (group/single-handed/number of practitioners/EMHS) will be requested as well.

Patient level

Outcomes:

All data will be extracted from the EHR of the general practitioner for all patients who satisfy the eligibility criteria. Data will be extracted at baseline and after 6 months. First, at baseline and after 6 months, all patients with a registered diagnosis of HF will be identified in the EMHS. Demographic data can be extracted with an automated search; other data will need to be collected by manual chart review. Additionally, all identified HF patients will be visited by the HF nurse at baseline and after 6 months and will be asked to fill in the MLHF-Q. At this occasion grip strength will be measured in the dominant hand using a JAMAR® Plus digital hand-held dynamometer. Three attempts at maximal squeeze will be recorded.

Process evaluation:

GPs will be asked to fill in a study registration form about the indication and results of their NT-proBNP POC test use and how it influenced their decision-making. The HF nurse will keep a log of all actions. Consequence of these actions will be collected from the patients' medical record. GPs will be asked to take note of the HF nurse advice in the EHR and indicate if it influenced decision-making.

Experiences of GPs and investigators:

The feedback meeting at 6 months will be organized as a focus group in each GP practice to get more insight in the experiences of the participating physicians and investigators. The meetings will be audiotaped and typed out. Any harm as a result of the trial will be explicitly collected and reported.

Practice level

Impact of the intervention on hospitalizations and mortality cannot be studied in this pilot trial, however, in a later stage this would be the outcome in the larger cluster-randomized trial, therefore, the feasibility of collecting data on hospitalizations and mortality will be tested. These outcomes will be measured at practice level in all patients aged 40 years or older, enlisted in one of the participating GP practices. GPs will be asked to register date of death and cause of death in the EHR of all patients who die during the study course. A list of hospitalized patients of each participating GP will be collected in all the surrounding hospitals (ZOL Genk, AZ Vesalius, Jessa Hasselt) and handed over to the GPs. Cause of hospitalization will be deducted from the discharge letter in the EHR by the GP in a standardized manner (trained by principal investigator (PI)). The anonymized data will be handed over to the PI.

Data management:

Data collection and data entries will be done by the PI and an assisting data manager. All patient data will be coded and anonymized. All other authors will have full access to the coded data (including statistical reports and tables) in the study and will be able to take responsibility for the integrity of the data and the accuracy of the data analysis.

Data analysis:

Descriptive statistics will be provided regarding baseline variables of the HF patients and general practitioners/general practices. Outcomes measured before and after the study intervention will be compared with a chi-squared test. Experiences of participating GPs and investigators will be analyzed qualitatively using thematic analysis as method.

Ethics:

Before the study start the investigators will present the participating physicians with an informed consent that outlines the intervention and the purpose of the trial. Additionally, all identified HF patients will be visited by the HF nurse before the start of the study. On that occasion the HF nurse will inform all HF patients about the study outline and purpose and ask informed consent. Furthermore, patients eligible for a NT-proBNP POC test will be informed by their GPs about the study outline and purpose and asked informed consent. However, informed consent cannot be sought for all patients on practice level (hospitalizations/mortality). Therefore, information about the study intervention and purpose of the trial will be presented on a poster in each practice, visible for all patients, who can opt-out if they object to study participation.

ELIGIBILITY:
Inclusion Criteria:

Heart failure patients are included if:

* They have their electronic medical records ("globaal medisch dossier") registered with one of the participating general practitioners.
* They have a registered diagnosis of HF (ICPC-2 code K77 or free text) in their electronic health record (EHR).

Patients can be included during the study if:

* They give their informed consent to participate in the study.
* Are eligible for a NT-proBNP POC test.

Exclusion Criteria:

* No exclusion criteria will be set

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the use of NT-proBNP POC test | 6 months
  How often do GPs use the POC test, for which indications, influence on decision-making?
Evaluation of the use of specialized HF nurse assistance | 6 months
  How often and for which indications do GPs use the assistance of the specialized HF nurse?

SECONDARY OUTCOMES:
Adequacy of HF diagnosis | 6 months
  Number of registered HF patients. Number of registered HF patients referred for echocardiography.
Adequacy of HF treatment | 6 months
  Number of HFrEF patients treated with RAAS-blockade, B-blockers or MRAs. The number of HFrEF patients treated with RAAS-blockade/B-blockers with a dose higher than starting dose
Evolution of HF patients' QoL | 6 months
  Evolution in quality of life of HF patients measured with a validated dutch version of the Minnesota living with heart failure questionnaire
Number of hospitalizations (all-cause, cardiovascular, HF-related) | 6 months
  the number of patients that are hospitalized at practice level
Mortality (all-cause/cardiovascular) | 6 months
  the number of patients that die during study course at practice level
Adequacy of follow-up | 6 months
  The number of HF patients that consulted their GP in the past 6 months
Adequacy of specialized follow-up | 6 months
  The number of HF patients that were referred to a cardiologist in the past 18 months
Adequacy of transition of care | 6 months
  The number of patients that contacted a familiar physician (cardiologist, GP, HF nurse) in the first 30 days after hospitalization

OTHER OUTCOMES:
Experiences of GPs with a multifaceted intervention to optimize care | 6 months
  Is a multifaceted intervention to optimize care feasible? How do GPs experience such an intervention?

CONTACTS AND LOCATIONS:
Overall Officials: Bert Aertgeerts, MD, PhD, Principal Investigator — Department of Public Health and Primary Care
Locations (1):
- Departement of Public Health and Primary Care, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smeets M, Raat W, Aertgeerts B, Penders J, Vercammen J, Droogne W, Mullens W, Janssens S, Vaes B. Mixed-methods evaluation of a multifaceted heart failure intervention in general practice: the OSCAR-HF pilot study. ESC Heart Fail. 2023 Apr;10(2):907-916. doi: 10.1002/ehf2.14251. Epub 2022 Dec 3. PMID 36461750